CLINICAL TRIAL: NCT05389267
Title: Safety Assessment of T4090 Eye Drops in Ocular Hypertensive or Glaucomatous Patients.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT4090-101
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T4090 (Experimental)
  Interventions: Drug: Kinezodianone R hydrochloride
- Placebo (Placebo Comparator): named "Vehicle" in the study protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kinezodianone R hydrochloride — Eyedrops
  Arms: T4090
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study purpose is to evaluate the safety of T4090.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent dated and signed.
* Both eyes diagnosed open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* History of trauma, infection, clinically significant inflammation within the previous 6 months
* Known or suspected hypersensitivity to one of the components of the Investigational Medicinal Product(s)
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ocular and systemic adverse events | up to 22 days
  Ocular and systemic treatment-emergent adverse events, serious TEAE, IMP-related TEAE, TEAE leading to premature IMP discontinuation.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr EL-HARAZI, Glendale, California, United States